CLINICAL TRIAL: NCT02053714
Title: Improving Diabetes Outcomes for Persons With Severe Mental Illness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: North Carolina Translational and Clinical Sciences Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 13-3211
Record Dates: First submitted 2014-01-21; First posted 2014-02-04 (Estimated); Last update posted 2017-05-09 (Actual); Status verified 2016-05

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus | interventions — Educational Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Self-management and education group (Other): Self-management and education group - 8 weeks of group-based information and activities designed to improve diabetes self-management
  Interventions: Behavioral: Diabetes self-management and education

INTERVENTIONS:
Behavioral: Diabetes self-management and education

SUMMARY:
Persons with severe mental illness are at great risk for developing type 2 diabetes (T2DM). Unfortunately, persons with mental illness and T2DM are less likely to receive recommended diabetes monitoring and are more likely to have poorly controlled diabetes, which leads to microvascular and macrovascular complications later in life. Evidence-based diabetes self-management education and support interventions have yet to be adapted for persons with mental illness and there have been no randomized controlled trials (RCTs) to examine their feasibility and efficacy. The purpose of this study is to assess the feasibility of conducting a RCT of a diabetes self-management intervention for persons with severe mental illness and T2DM.

ELIGIBILITY:
Inclusion Criteria: Type 2 diabetes plus severe mental illness -

Exclusion Criteria: None

-

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2013-12; Primary Completion 2015-06-15 (Actual); Study Completion 2015-12-31 (Actual)

PRIMARY OUTCOMES:
Changes in knowledge of diabetes self-management from baseline to six months as evidenced by scores on the Stanford Diabetes Self-Management Questionnaire. | Baseline, 6 months

SECONDARY OUTCOMES:
Changes in HBA1c values from baseline to six months. | Baseline, 6 months
Changes in diabetes self-efficacy from baseline to six months as evidenced by scores on the Stanford Diabetes Self-Efficacy Questionnaire. | Baseline, 6 months
Changes in eating self-efficacy from baseline to six months as evidenced by scores on a standardized measure of eating self-efficacy. | Baseline, 6 months
  Glynn and Ruderman's (1986) eating self-efficacy scale will be used.
  Glynn, S.M., & Ruderman, J. (1986). The development and validation of an eating self-efficacy scale. Cognitive Therapy and Research, 10, 403-420.
Changes in exercise self-efficacy from baseline to six months as evidenced by scores on a standardized measure of exercise self-efficacy. | Baseline, 6 months
  Bandura's exercise self-efficacy scale will be used. Bandura, A. (1997). Self-efficacy: The exercise of control. New York: W.H. Freeman.
Changes in healthy lifestyle activities from baseline to six months as evidenced by scores on a standardized measure of adult health behavior. | Baseline, 6 months
Changes in health promoting activities from baseline to six months as evidenced by scores on a standardized measure of health promoting lifestyle activities. | Baseline, 6 months
Changes in waist circumference from baseline to six months. | Baseline, 6 months
Changes in triceps circumference from baseline to six months. | Baseline, 6 months
Changes in subscapular skinfold measurement from baseline to 6 months. | Baseline, 6 months
Changes in body mass index from baseline to six months. | Baseline, 6 months
Changes in diastolic and systolic blood pressure from baseline to six months. | Baseline, 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Gary S Cuddeback, Ph.D., Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No